CLINICAL TRIAL: NCT06485856
Title: Cukurova University
Brief Title: ASSESSMENT OF PAIN USING A PAIN DIAGNOSTIC SYSTEM THAT MEASURS FACIAL MOVEMENT USING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatmagül Üstünel (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Sponsor-Investigator, Fatmagül Üstünel, Principal Investigator, Cukurova University
Organization: Cukurova University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FU312
Record Dates: First submitted 2024-06-06; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Nursing; Pain Assessment; Critical Care; Technology; Facial Recognition
Keywords: Nurse; Pain assessment; Intensive care; Facial diagnosis; Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Other): During the procedural procedures applied to patients who are monitored in intensive care and who are conscious but unable to express themselves verbally, their pictures will be taken 12 times for one minute. This procedure will be applied to the same patient during 4 different procedures. After the procedure, the patient will be asked to score his/her pain numerically between 0-10 (0-no pain, 10-severe/unbearable pain). In addition, the images obtained will be evaluated by three expert nurses and they will be asked to estimate the patient's pain based on their facial expressions. Meanwhile, the pain assessment based on the patient's pictures will be evaluated numerically between 0-10 by the Facial Action Coding system. As the final process, all data will be compared and the patient's pain expression will be compared with the Facial Action Coding system and the pain evaluations of the experts. The assessment closest to the patient's pain expression will be determined.
  Interventions: Behavioral: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

INTERVENTIONS:
Behavioral: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 — Evaluation of the pain level of patients who are followed in intensive care and cannot speak during the procedural procedure with 3 different methods.

SUMMARY:
Pain is a subjectively difficult, abstract and comprehensive concept that is at the core of the whole study, emerging in relation to various advancements, and detailed description. For non-controlling, stress-free, stress-or-thickness training for thromboembolic, pulmonary and other organ modalities, re-admission from discharge, thromboembolic, pulmonary and other reasons.

The scales of use in the assessment of pain in the conscious surgical patient who cannot communicate verbally, into the pain, are physically subjective. Ekman and Friesen are planning the movements of their muscles to be performed by an Action Coding process that could be experienced in 1978. system; It has been applied in pain, in the evaluation of pain in the postoperative period and in children, in the new clinical practice, and in the new and clinical practice.

Health professionals may be biased in diagnosing pain, especially in intensive care patients, and may underestimate pain. In the literature, it is seen that the child who is made with pain in his patients in education in the field of medicine is not used in his experiences, similar to the pain that measures the tastes of the faces of the single scales. In this context, standardized, continuous, objective and scalable pain measures indicate the practice environment. The aim of these people is to evaluate the pain in our surgical patients who cannot communicate clearly and clearly with pain diagnosis that measures facial movement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Those with intubation/tracheostomy,
* Conscious, unable to communicate verbally,
* Glaskow coma score 13-15,
* Patients who agreed to participate in the study

Exclusion Criteria:

* Those with any facial abnormality that may alter facial expression analysis (facial paralysis, Poland-mobius syndrome)
* Those with neurological and mental disorders,
* Having a history of chronic pain,
* Those who have a condition that requires them to be in the prone position all the time (Pilonidal Sinus, ARDS, etc.),
* Patients who cannot speak the same language as the healthcare professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Pain diagnosis in intensive care patients | In the intensive care unit, the pain felt by the patient during the procedure will be evaluated. This assessment will be repeated for each patient throughout the 12 procedure procedures performed on the patient.
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Cukurova University Cukurova University, Study Director — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)